CLINICAL TRIAL: NCT05989217
Title: Conservative Therapies in the Treatment of Temporomandibular Disorders: a Randomized Controlled Clinical Trial.
Brief Title: Conservative Therapies in the Treatment of Temporomandibular Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Alfenas (Other)
Responsible Party: Principal Investigator, Daniel Augusto de Faria Almeida, Principal Investigator, Universidade Federal de Alfenas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMJ Disorders
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Joint Pain; Splints; Photobiomodulation
Keywords: Temporomandibular Joint Disorders; Splints; Laser therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Occlusal Splints; Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Occlusal Splint (Experimental): Participants allocated will receive therapy with a stabilizing plate made by the simplified technique. This plate is made of an acetate plate, plasticized in a plaster model, and individualized by acrylic resin. This technique allows the professional to make and install the plate in a short time, without the laboratory step, and is also more economical.
  After the plate installation and adjustments, the participant will be instructed to use the device every night during sleep. Weekly adjustments will be performed for 4 weeks, and in these sessions information regarding the research parameters will be collected.
  Interventions: Device: Occlusal Splint
- Laser Therapy (Experimental): All participants will be examined and pain trigger points will be identified, if any. The laser will be applied at predetermined points and at specific trigger points identified during the clinical examination. The application of the laser will be symmetrical, i.e. on both sides of the face, with the same number of points, regardless of whether it is a "trigger point" or not.
  The equipment to be used and the parameters for the applications have the following characteristics: 808 nm wavelength, 100 mW of useful emitter power, 105 J/cm2 of energy density, spot area 0.028 cm2, Energy/point 3 J, 1 application per week for 4 weeks.
  Interventions: Radiation: Laser Therapy
- Occlusal Splint + Laser Therapy (Experimental): The therapies will be associated during the same period as the other groups, ensuring the same application and evaluation protocols.
  Interventions: Device: Occlusal Splint; Radiation: Laser Therapy
- Acupuncture Laser Therapy (Experimental): The laser will be applied to predetermined acupuncture points and specific trigger points identified during the clinical examination. The application will be performed symmetrically and bilaterally, regardless of the presence of trigger points. A standardized protocol will be followed for all participants, irrespective of tissue thickness or gender. The equipment to be used will emit an infrared light beam with a wavelength of 808 nm, output power of 100 mW, energy density of 105 J/cm², and a spot size of 0.028 cm², delivering 3 J per point, which corresponds to a 30-second application per point. The protocol will consist of five applications: one at baseline, followed by four weekly sessions.
  Interventions: Radiation: Acupuncture Laser Therapy
- Occlusal Splint + Acupuncture Laser Therapy (Experimental): In the combined therapy group, the therapies will be administered simultaneously with those of the other groups, ensuring standardized protocols for application and evaluation throughout the study period.
  Interventions: Device: Occlusal Splint; Radiation: Acupuncture Laser Therapy

INTERVENTIONS:
Device: Occlusal Splint — Occlusion Splint
  Arms: Occlusal Splint; Occlusal Splint + Acupuncture Laser Therapy; Occlusal Splint + Laser Therapy
Radiation: Laser Therapy — Laser Therapy
  Arms: Laser Therapy; Occlusal Splint + Laser Therapy
Radiation: Acupuncture Laser Therapy — Acupuncture Laser Therapy
  Arms: Acupuncture Laser Therapy; Occlusal Splint + Acupuncture Laser Therapy

SUMMARY:
The present study was designed to evaluate different conservative therapies in patients with temporomandibular disorders. A total of 160 patients will be selected after the diagnosis of TMD according to the Diagnostic Criteria for Temporomandibular Disorder (DC/TMD), axis I. Patients will be randomly divided into five groups: OD group (n=32): treated with an occlusal device; LLLT group (n=32): treated with infrared low-level laser; ODL group (n=32): treated with OD + LLLT; LAT group (n=32): treated with laser acupuncture and ODLAT group (n=32): treated with both OD and LAT. Patients undergoing therapy with a stabilizing plate (made using the simplified technique) will be instructed to use the device every night while sleeping for four weeks. In both the LLLT and LAT groups, the protocol involved five applications: one at baseline, followed by four subsequent weekly sessions. The intensity of pain will be classified using the Visual Analog Scale (VAS). Mandible function will be assessed by maximum unassisted mouth opening. The impact of therapies on oral health will also be evaluated using the Oral Health Impact Profile (OHIP-14) instrument in a simplified form.

ELIGIBILITY:
Inclusion Criteria:

* Adults of legal age
* Both sexes
* Regardless of race or social class
* With the main complaint of pain in the temporomandibular joint or orofacial region
* With or without limitation of mouth opening, diagnosed through the DC/TMD axis1, with pain in the masticatory mm and muscular TMD
* Participants must have complete permanent dentition and normal occlusion.

Exclusion Criteria:

* Congenital problems affecting the TMJ and/or orofacial and cervical region of the skull;
* Neoplastic conditions;
* History of recent trauma to the orofacial/cervical region of the skull;
* Previous use of any type of TMD treatment plate;
* Current use of functional orthopedic appliances or fixed and/or removable orthodontic appliances;
* Cleft lip and/or palate syndromes;
* Psychiatric disorders;
* Severe cardiac problems;
* A severely poor dental condition such as periodontitis and/or indication for endodontic treatment;
* Those using topical or systemic photosensitizing drugs;
* Pregnant women;
* Dermatological diseases in the region where irradiation will be performed;
* Patients with impaired cognitive ability;
* History of head trauma related to the etiology of orofacial pain;
* Migraine or intracranial disorders;
* Who used medications in the last 3 months that may interfere with the effect of therapies, such as relaxants, anticonvulsants and who used medications to treat TMD or muscular pain;
* Who had other causes of orofacial pain, such as caries, neuropathies and fibromyalgia;
* Who had phobia about needles or bleeding disorders;
* Patients who are unable to attend the clinic during the prescribed treatment period;
* Patient who insists on a specific treatment (e.g. occlusal adjustments, medication);
* Presence of removable full or partial dentures with distal extension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain in the Temporomandibular Joint and/or masticatory muscles | Change from baseline pain at 0, 1, 2, 3, 4 and 12 weeks.
  The visual analog scale (VAS) will be used to quantify spontaneous pain in the Temporomandibular Joint and/or masticatory muscles at rest or during palpation. The VAS is a line (ruler) 10 cm long, with a left end point indicating a pain-free state and a right end point indicating the greatest imaginable pain.

SECONDARY OUTCOMES:
Mouth opening | Change from baseline mouth opening at 0, 1, 2, 3, 4, and 12 weeks.
  Pain-free opening is defined as the maximum amount a patient can achieve when opening their mouth without experiencing pain and will be measured as the distance between the incisal edges of the upper and lower central incisors.
  Maximum unassisted mouth opening will be measured as the distance between the upper and lower central incisors and defined as the greatest amount of opening a patient can achieve regardless of pain and discomfort.
Oral Health Impact Profile | Change from baseline Oral Health Impact Profile at 0, 5 and 12 weeks.
  The impact of oral health-related quality of life will be analyzed using the Oral Health Impact Profile - Short form (OHIP-14) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Almeida, PhD, Principal Investigator — Universidade Federal de Alfenas
Locations (1):
- Universidade Federal de Alfenas, Alfenas, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No